CLINICAL TRIAL: NCT04432181
Title: Associated Professor, Director of Strabismus Department
Brief Title: Comparison of Deviation Types Among Astigmatic Children With Or Without Amblyopia
Status: Completed | Type: Observational
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, Burçin Çakır, Burcin Cakir, FICO, Sakarya University
Other Study IDs: sakarya amblyopia
Record Dates: First submitted 2020-06-11; First posted 2020-06-16 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Astigmatism of Both Eyes; Amblyopia; Strabismus
MeSH Terms: conditions — Amblyopia; Strabismus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1, astigmatic patients with amblyopia: astigmatic children with amblyopia
  Interventions: Other: ophthalmic examination
- Group 2, astigmatic patients without amblyopia: astigmatic children without amblyopia
  Interventions: Other: ophthalmic examination

INTERVENTIONS:
Other: ophthalmic examination — ophthalmic examination including; best corrected visual acuity, alternating prism cover test, retinoscopy, fundus examination, ocular vergence evaluation

SUMMARY:
the records of astigmatic children were reviewed and any deviation was investigated at near and distance. refractive errors, stereopsis, convergence insufficiency were also evaluated. children were divided into two groups according to the presence of amblyopia and ocular deviations and other parameters were compared between groups.

DETAILED DESCRIPTION:
The aim of the study was to evaluate deviations in children with ≥1,75 diopter (D) astigmatism with or without amblyopia.

The records of children with ≥1,75 D astigmatism were investigated. Subjects with and without amblyopia composed group 1 and 2, respectively. The mean age, gender, amount and type of deviation, presence of convergence insufficiency (CI), stereopsis, time of initial spectacle use and follow-up time, differences in best corrected visual acuity (VoD) and spherical equivalent (SE) between eyes were noted and compared between the groups. Best corrected visual acuity (BCVA), mean SE, astigmatism measurements were also noted and compared between amblyopic, fellow and non-amblyopic eyes.

ELIGIBILITY:
Inclusion Criteria:

* astigmatisma ≥1,75 Diopter

Exclusion Criteria:

* systemic diseases additional ocular diseases neurological diseases

Ages: 7 Years to 13 Years | Sex: All
Age Groups: Child
Study Population: children age range between 7 and 13 years with ≥1,75 diopter (D) astigmatism were included. Patients with additional ocular and systemic diseases were excluded in this study. Subjects with and without amblyopia composed group 1 and 2, respectively.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2018-09-04 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2020-02-03 (Actual)

PRIMARY OUTCOMES:
ocular deviation | 24 month
  ocular deviation measured by alternate prism cover test, prism diopter

SECONDARY OUTCOMES:
convergence | 24 month
  presence of convergence insufficiency at 10 cm far from visual axe.

CONTACTS AND LOCATIONS:
Overall Officials: Burcin Cakir, MD, Principal Investigator — Sakarya University
Locations (1):
- Sakarya University Ophthalmology Department, Sakarya, Turkey (Türkiye)